CLINICAL TRIAL: NCT05658692
Title: Platform Adaptive Embedded Trial for Acute Respiratory Distress Syndrome
Acronym: PETARDS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); West China Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Peking Union Medical College Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fudan University (Other); Guangdong Provincial People's Hospital (Other); Ningbo No. 1 Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0770
Record Dates: First submitted 2022-11-22; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; ICU; domain; platform adaptive embedded trial
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Dexamethasone; Hydrocortisone; 3-hydroxyphenyltrimethylammonium; Vecuronium Bromide; Succinylcholine; Simvastatin; Rosuvastatin Calcium; Extracorporeal Membrane Oxygenation; Propofol; Midazolam; Dexmedetomidine; Dopamine; olprinone; Simendan; Norepinephrine; Epinephrine; Metaraminol; Isoproterenol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- protective ventilation (Experimental): For ARDS patients with moderate to severe mechanical ventilation(MAQUET), give 6-8ml/kg (ideal body weight PBW), and control the plateau pressure to <30cmH2O; In patients with respiratory distress, the tidal volume can be increased to 7-8ml/kg (PBW), while the plateau pressure is <30cmH2O. Adjust breathing rate according to CO2 level, up to 35 breaths/min. PBW, male: 50+0.91 (height cm-152.4); female: 45.5+0.91 (height cm-152.4).
  Interventions: Device: protective ventilation
- prone position ventilation (including awake state) (Experimental): For patients with moderate to severe ARDS who have no contraindications to prone ventilation, protective lung ventilation is given and prone ventilation is performed; the duration is more than 12 hours/time.
  Interventions: Behavioral: prone position ventilation
- glucocorticoid therapy (Experimental): Glucocorticoids are used for ARDS patients, with small doses and short courses of treatment in the acute phase (within 14 days). There is no clear recommendation for patients with ARDS from other causes. At present, the main research methods are methylprednisolone program(Solu-Medrol®), dexamethasone program, and hydrocortisone program
  Interventions: Drug: glucocorticoid therapy
- restrictive fluid resuscitation (Experimental): ARDS patients with circulatory or organ hypoperfusion problems should use as little fluid as possible to maintain treatment and circulation; other ARDS patients should focus on stabilizing circulation during the resuscitation phase, with controlled fluid replacement combined with early vasoactive drugs; ultrasound, Central venous pressure measurement, mixed central venous oxygen saturation, alveolar-arterial oxygen difference, blood lactate, etc. guide fluid resuscitation therapy; stop using vasoactive drugs for more than 12 hours, and use diuretics or diuretics combined with albumin to achieve fluid balance.
  Interventions: Other: restrictive fluid resuscitation
- Immunomodulatory therapy (Experimental): Thymosin Alpha（Thymalfasin for Injection） 1.6mg subcutaneously twice a week.
  Interventions: Biological: Thymosin Alpha
- Muscle relaxant therapy (Experimental): For patients with moderate to severe ARDS, if light sedation cannot achieve protective lung ventilation strategy and prone position ventilation, deep sedation combined with intermittent bolus injection of muscle relaxants（Vecuronium Bromide for Injection） is used; if protective lung ventilation strategy and prone position ventilation still cannot be achieved, deep sedation combined with continuous Inject muscle relaxants.
  Interventions: Drug: Muscle relaxant therapy
- Integrated Chinese and Western Medicine Treatment (Experimental): Mechanical ventilation + conventional western medicine + Dachengqi Decoction/Rhubarb-Salvia Injection/Tanreqing/Xuanbai Chengqi Decoction(Drugs determined by syndrome differentiation and treatment)
  Interventions: Other: Integrated Chinese and Western Medicine Treatment
- statin therapy (Experimental): There are currently two options: 1) Simvastatin （Simvastatin Tablets）80 mg QD orally for up to 28 days in patients with acute lung injury. 2) Rosuvastatin （Rosuvastatin Calcium Tablets）40 mg for the first time, followed by 20 mg orally daily for 28 days, or 3 days after being transferred out of the ICU, or after the patient died.
  Interventions: Drug: statin therapy
- anti-infective treatment (Experimental): Refer to the "Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021." recommendations.
  Interventions: Combination Product: anti-infective treatment
- Extracorporeal Membrane Oxygenation（ECMO） (Experimental): ECMO (Medtronic) is chosen as rescue therapy for severe ARDS patients with refractory hypoxemia within 7 days of onset. (Oxygenation index < 50 mmHg for 3 hours, or oxygenation index < 80 mmHg for 6 hours, or arterial pH < 7.25, arterial partial pressure of carbon dioxide [Paco2] ≥ 60 mmHg > 6 hours, and respiratory rate increased to every minute 35 breaths, adjusting mechanical ventilation settings to maintain plateau pressure ≤32 cmH2O) despite ventilator optimization (defined as inspired oxygen concentration) ≥ 0.80, tidal volume 6 ml/kg (PBW), and positive end-expiratory pressure [PEEP] ≥ 10 cmH2O). V-V mode is preferred.
  Interventions: Device: Extracorporeal Membrane Oxygenation（ECMO）
- stem cell therapy (Experimental): Previous clinical studies have found that stem cell therapy is safe, using a single injection of bone marrow stem cells at a dose of 1, 5, 10*106 cells/kg; START trial, ClinicalTrials.gov NCT02097641, for patients with moderate to severe ARDS, a single intravenous injection of bone marrow stem cells 10* 106 cells/kg intervention protocol.
  Interventions: Genetic: stem cell therapy
- Sedative analgesia/muscle relaxant therapy (Experimental): For patients with moderate to severe ARDS, if light sedation cannot achieve protective lung ventilation strategy and prone position ventilation, deep sedation（Propofol Injectable Emulsion or Midazolam Injection） combined with intermittent bolus injection of muscle relaxants is used; if protective lung ventilation strategy and prone position ventilation still cannot be achieved, deep sedation combined with continuous Inject muscle relaxants（Vecuronium Bromide for Injection）.
  Interventions: Drug: Sedative analgesia/muscle relaxant therapy
- inotropes therapy (Experimental): For unconventional medication, according to"Surviving sepsis campaign: international guidelines for the management of sepsis and septic shock 2021".
  Interventions: Drug: inotropes therapy
- Vasoactive drug therapy (Experimental): According to"Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021".
  Interventions: Drug: Vasoactive drug therapy

INTERVENTIONS:
Device: protective ventilation — Patients with moderate to severe ARDS received ventilation treatment according to predicted body weight(PBW) and controlled plateau pressure.
  Arms: protective ventilation
Behavioral: prone position ventilation — patients with moderate to severe ARDS who don't have contraindications were given prone ventilation for over 12 hours.
  Arms: prone position ventilation (including awake state)
Drug: glucocorticoid therapy — Dexamethasone: Patients received intravenous dexamethasone 20 mg daily from days 1 to 5, reduced to 10 mg daily from days 6 to 10.
  Hydrocortisone：For septic ARDS patients, 50 mg of hydrocortisone was given as an intravenous bolus every 6 hours for 7 days; For patients with COVID-19-related ARDS, The corticosteroid field randomized participants to a fixed 7-day period of intravenous hydrocortisone (50 mg or 100 mg every 6 hours).
  Other Names: Dexamethasone; Hydrocortisone
  Arms: glucocorticoid therapy
Other: restrictive fluid resuscitation — 1. without other organ dysfunction patients: Minimize fluid was given;
  2. other ARDS patients: In the resuscitation phase, controlled fluid replacement combined with vasoactive drugs was given; multiple measures were taken, like lactate and so on, to utilizedto guide fluid resuscitation therapy; diuretics or diuretics in combination with albumin to achieve fluid balance.
  Arms: restrictive fluid resuscitation
Biological: Thymosin Alpha — People received thymosin Alpha subcutaneous injections, twice a week.
  Arms: Immunomodulatory therapy
Drug: Muscle relaxant therapy — Deep sedation combined with intermittent bolus injection of muscle relaxant or deep sedation combined with continuous infusion of muscle relaxant
  Other Names: Vecuronium Bromide; Succinylcholine
  Arms: Muscle relaxant therapy
Other: Integrated Chinese and Western Medicine Treatment — 1. ventilation;
  2. conventional western medicine treatment；
  3. Chinese herbal medicine（Determining medication based on syndrome differentiation）
  Arms: Integrated Chinese and Western Medicine Treatment
Drug: statin therapy — 1. Simvastatin: 80mg qd po for not more than 28days;
  2. Rosuvastatin: 20mg qd po (40mg for the first time) for 28days or 3 days after transfer out of the ICU, or the patient died.
  Other Names: Simvastatin; Rosuvastatin
  Arms: statin therapy
Combination Product: anti-infective treatment — According to "Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021".
  Arms: anti-infective treatment
Device: Extracorporeal Membrane Oxygenation（ECMO） — 1. For severe ARDS patients with refractory hypoxemia within 7 days of onset;
  2. (Inspiratory oxygen concentration) ≥ 0.80, tidal volume 6ml/kg (PBW), positive end-expiratory pressure [PEEP] ≥ 10 cmH2O;
  3. V-V Model.
  Arms: Extracorporeal Membrane Oxygenation（ECMO）
Genetic: stem cell therapy — A single injection of bone marrow stem cells, doses of 1, 5, 10*106 cells/kg was taken according to the previous clinical studies.
  Arms: stem cell therapy
Drug: Sedative analgesia/muscle relaxant therapy — Deep sedation combined with intermittent bolus injection of muscle relaxant or deep sedation combined with continuous infusion of muscle relaxant
  Other Names: Propofol; midazolam; dexmedetomidine
  Arms: Sedative analgesia/muscle relaxant therapy
Drug: inotropes therapy — According to "Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021".
  Other Names: Dopamine; Olprinone; Levosimendan
  Arms: inotropes therapy
Drug: Vasoactive drug therapy — According to "Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021".
  Other Names: Norepinephrine; epinephrine; metaraminol; isoproterenol
  Arms: Vasoactive drug therapy

SUMMARY:
Platform adaptive embedded trial for acute respiratory distress syndrome (PETARDS) is a randomized, embedded, multifactorial, adaptive platform trial for ARDS. The study aimed to assess the impact of multiple interventions on outcomes in patients with ARDS admitted to the ICU.

DETAILED DESCRIPTION:
Mortality is significantly higher in ARDS patients requiring intensive care unit (ICU) admission.

ARDS patients admitted to the ICU typically receive multiple (as many as 10 or 20) treatments that work together to fight infection, reduce pulmonary exudation, improve oxygenation, and support systemic organ function. Clinicians are often willing to choose the exact or considered safe and effective regimen from the therapies mentioned above. Still, there are individual differences in ARDS patients, and it is difficult to confirm the optimal treatment plan. It is inevitable to choose treatment without evidence-based medicine based on experience. The primary purpose of this study was to help physicians select the best-effective approach among existing ARDS therapies, and secondly to provide a rationale for specific empirical or emerging ARDS treatments.

Clinical evidence to guide optimal management is best obtained from randomized controlled trials (RCTs); however, ARDS is a multi-causal, clinically and therapeutically heterogeneous clinical syndrome with rapid disease progression and complex clinical manifestations, in fact, difficult to organize RCT trials. In cases where the timing of onset and the pathophysiological mechanism cannot be determined, the initial treatment is the selection of protective ventilation/controlled infusion as the first-line standard therapy according to the Berlin classification of ARDS, and some second-line treatments with potential clinical benefit. It is difficult to conduct objective, scientific and timely evaluation, and the overall treatment plan is inevitably blind and empirical. This clinical operation mode is likely related to ARDS-related RCT research results. The results are unsatisfactory, the treatment response heterogeneity is high, and the outcome events vary greatly. closely related to the clinical status. The adaptive platform trial PETARDS is ideal for evaluating the effects of highly heterogeneous ARDS treatment strategies.

This clinical research design (adaptive platform trial, APT) can use the information of patients who are participating in the study to guide the clinical treatment of subsequent newly enrolled patients.

The APT trial randomized patients into multiple domains for multiple interventions to assess their effectiveness in different patients. The term "domain" refers to a common treatment unit (eg, steroid therapy) within which patients can be randomly assigned to several interventional (dose) groups (including controls, such as no steroids, as appropriate). Certainly). All trial procedures consist of a primary or "core" protocol and multiple secondary protocols, and the standard protocols, clinical treatment adaptations, and trial management and practices for specific treatment units are managed in a unified manner for each treatment unit. The core protocol, secondary protocols, and Statistical Analysis Plan (SAP) of this trial are presented in the appendix; the study required approval from the relevant ethics committees of all participating hospitals and was conducted by good clinical practice guidelines and principles described in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (18 years and older, regardless of gender) admitted to the ICU with ARDS; Intubation and mechanical ventilation; Moderate/severe ARDS defined by Berlin criteria (PaO2/FiO2 ≤200mmHg, PEEP ≥5cmH20); Moderate/severe ARDS less than 48 hours before randomization.

Exclusion Criteria:

Pregnancy or breastfeeding; Known allergy to the intervention drug; Daily use of an intervention drug or measure within the past 15 days; Intervention drugs or measures primarily intended to treat other conditions (eg, septic shock); Patients using the intervention drug or standard for two or more days during hospitalization; Patients are expected to die within the next 24 hours; Other: Participated in PETARDS in the past 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
ventilator-free days | within 28 days
  Ventilator-free days 28 days after randomization, definition: Survival without mechanical ventilation

SECONDARY OUTCOMES:
Clinical status assessment | 15 days
  Patients' clinical status (6-point scale score) was assessed on day 15 after randomization, Definition: This scale ranges from 1 (no hospitalization) to 6 (death), with higher scores indicating worse outcomes.
All-Cause Mortality | within 28 days
  All-cause mortality 28 days after randomization
Duration of mechanical ventilation | within 28 days
  days of mechanical ventilation
Sequential Organ Failure Assessment (SOFA) Score | at 48 hours, 72 hours, and 7 days after randomization
  SOFA Score for different times, from 0 to 24 points
ICU stay time | within 90 days
  The time for patients staying in ICU when they were in the hospital.
Hospital stay | within 90 days
  The whole time patients lived in the hospital, including the time when they lived in the ICU
Organ failure free days | within 28 days
  Patients got ARDS, but the other organs were not injury.
Health-related quality of life assessment, EQ5D-5L and WHODAS 2.0 | within 6 months
  Patient's life quality was assessed according to EQ5D-5L. If the patient had severe impairment of organ function within 6 months, evaluated the patient's quality of life according to WHODAS 2.0
Proportion of intubated patients undergoing tracheostomy | 28 days
  ARDS patients received tracheostomy.
Where the patient went after discharge | No recurrence within 90 days
  Home, rehabilitation hospital, nursing home or long-term care facility, or other emergency hospital
Re-admission to ICU during readmission | within 90 days
  Patients were sent to the hospital and sent to the ICU again,
Days not in intensive care unit | 28 days after randomization
  ICU transfer and discharge 28 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zhaocai Zhang, Doctor, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (11):
- China (11):
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital，Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangdong
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Lanxi People's Hospital, Lanxi
  - Ningbo First Hospital, Ningbo
  - Zhognshang hospital, Fudan University, Shanghai
  - Taizhou Hosptial of Zhejiang Province, Taizhou
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Wuhan University Renmin Hospital, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
1. all collected IPD；
  2. all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be permanently available after the publication of this study.
Access Criteria: Data will be made available to all upon publication of this study. Applicants can contact the corresponding author to apply, but they must provide the reasons for the application, the purpose of the research, and the ethical certificates of the relevant research.

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Annane D, Pastores SM, Rochwerg B, Arlt W, Balk RA, Beishuizen A, Briegel J, Carcillo J, Christ-Crain M, Cooper MS, Marik PE, Umberto Meduri G, Olsen KM, Rodgers S, Russell JA, Van den Berghe G. Guidelines for the diagnosis and management of critical illness-related corticosteroid insufficiency (CIRCI) in critically ill patients (Part I): Society of Critical Care Medicine (SCCM) and European Society of Intensive Care Medicine (ESICM) 2017. Intensive Care Med. 2017 Dec;43(12):1751-1763. doi: 10.1007/s00134-017-4919-5. Epub 2017 Sep 21. PMID 28940011
- [Background] Meduri GU, Annane D, Confalonieri M, Chrousos GP, Rochwerg B, Busby A, Ruaro B, Meibohm B. Pharmacological principles guiding prolonged glucocorticoid treatment in ARDS. Intensive Care Med. 2020 Dec;46(12):2284-2296. doi: 10.1007/s00134-020-06289-8. Epub 2020 Nov 4. PMID 33150472
- [Background] Villar J, Ferrando C, Martinez D, Ambros A, Munoz T, Soler JA, Aguilar G, Alba F, Gonzalez-Higueras E, Conesa LA, Martin-Rodriguez C, Diaz-Dominguez FJ, Serna-Grande P, Rivas R, Ferreres J, Belda J, Capilla L, Tallet A, Anon JM, Fernandez RL, Gonzalez-Martin JM; dexamethasone in ARDS network. Dexamethasone treatment for the acute respiratory distress syndrome: a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Mar;8(3):267-276. doi: 10.1016/S2213-2600(19)30417-5. Epub 2020 Feb 7. PMID 32043986
- [Background] Vignon P, Evrard B, Asfar P, Busana M, Calfee CS, Coppola S, Demiselle J, Geri G, Jozwiak M, Martin GS, Gattinoni L, Chiumello D. Fluid administration and monitoring in ARDS: which management? Intensive Care Med. 2020 Dec;46(12):2252-2264. doi: 10.1007/s00134-020-06310-0. Epub 2020 Nov 9. PMID 33169217
- [Background] Malbrain MLNG, Van Regenmortel N, Saugel B, De Tavernier B, Van Gaal PJ, Joannes-Boyau O, Teboul JL, Rice TW, Mythen M, Monnet X. Principles of fluid management and stewardship in septic shock: it is time to consider the four D's and the four phases of fluid therapy. Ann Intensive Care. 2018 May 22;8(1):66. doi: 10.1186/s13613-018-0402-x. PMID 29789983
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Alhazzani W, Belley-Cote E, Moller MH, Angus DC, Papazian L, Arabi YM, Citerio G, Connolly B, Denehy L, Fox-Robichaud A, Hough CL, Laake JH, Machado FR, Ostermann M, Piraino T, Sharif S, Szczeklik W, Young PJ, Gouskos A, Kiedrowski K, Burns KEA. Neuromuscular blockade in patients with ARDS: a rapid practice guideline. Intensive Care Med. 2020 Nov;46(11):1977-1986. doi: 10.1007/s00134-020-06227-8. Epub 2020 Oct 26. PMID 33104824
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] McAuley DF, Laffey JG, O'Kane CM, Cross M, Perkins GD, Murphy L, McNally C, Crealey G, Stevenson M; HARP-2 investigators; Irish Critical Care Trials Group. Hydroxymethylglutaryl-CoA reductase inhibition with simvastatin in acute lung injury to reduce pulmonary dysfunction (HARP-2) trial: study protocol for a randomized controlled trial. Trials. 2012 Sep 17;13:170. doi: 10.1186/1745-6215-13-170. PMID 22985805
- [Background] McAuley DF, Laffey JG, O'Kane CM, Perkins GD, Mullan B, Trinder TJ, Johnston P, Hopkins PA, Johnston AJ, McDowell C, McNally C; HARP-2 Investigators; Irish Critical Care Trials Group. Simvastatin in the acute respiratory distress syndrome. N Engl J Med. 2014 Oct 30;371(18):1695-703. doi: 10.1056/NEJMoa1403285. Epub 2014 Sep 30. PMID 25268516
- [Background] National Heart, Lung, and Blood Institute ARDS Clinical Trials Network; Truwit JD, Bernard GR, Steingrub J, Matthay MA, Liu KD, Albertson TE, Brower RG, Shanholtz C, Rock P, Douglas IS, deBoisblanc BP, Hough CL, Hite RD, Thompson BT. Rosuvastatin for sepsis-associated acute respiratory distress syndrome. N Engl J Med. 2014 Jun 5;370(23):2191-200. doi: 10.1056/NEJMoa1401520. Epub 2014 May 18. PMID 24835849
- [Background] Combes A, Hajage D, Capellier G, Demoule A, Lavoue S, Guervilly C, Da Silva D, Zafrani L, Tirot P, Veber B, Maury E, Levy B, Cohen Y, Richard C, Kalfon P, Bouadma L, Mehdaoui H, Beduneau G, Lebreton G, Brochard L, Ferguson ND, Fan E, Slutsky AS, Brodie D, Mercat A; EOLIA Trial Group, REVA, and ECMONet. Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome. N Engl J Med. 2018 May 24;378(21):1965-1975. doi: 10.1056/NEJMoa1800385. PMID 29791822
- [Background] Brodie D, Bacchetta M. Extracorporeal membrane oxygenation for ARDS in adults. N Engl J Med. 2011 Nov 17;365(20):1905-14. doi: 10.1056/NEJMct1103720. PMID 22087681
- [Background] Qin H, Zhao A. Mesenchymal stem cell therapy for acute respiratory distress syndrome: from basic to clinics. Protein Cell. 2020 Oct;11(10):707-722. doi: 10.1007/s13238-020-00738-2. Epub 2020 Jun 9. PMID 32519302
- [Background] Matthay MA, Calfee CS, Zhuo H, Thompson BT, Wilson JG, Levitt JE, Rogers AJ, Gotts JE, Wiener-Kronish JP, Bajwa EK, Donahoe MP, McVerry BJ, Ortiz LA, Exline M, Christman JW, Abbott J, Delucchi KL, Caballero L, McMillan M, McKenna DH, Liu KD. Treatment with allogeneic mesenchymal stromal cells for moderate to severe acute respiratory distress syndrome (START study): a randomised phase 2a safety trial. Lancet Respir Med. 2019 Feb;7(2):154-162. doi: 10.1016/S2213-2600(18)30418-1. Epub 2018 Nov 16. PMID 30455077
- [Background] Wick KD, Leligdowicz A, Zhuo H, Ware LB, Matthay MA. Mesenchymal stromal cells reduce evidence of lung injury in patients with ARDS. JCI Insight. 2021 Jun 22;6(12):e148983. doi: 10.1172/jci.insight.148983. PMID 33974564